CLINICAL TRIAL: NCT03710395
Title: Influence of Genetic Polymorphisms of ABCG2/BCRP on the Transport of Nifedipine to Breast Milk in Hypertensive Breastfeeding Women.
Brief Title: Genetic Polymorphisms of ABCG2/BCRP on the Transport of Nifedipine to Breast Milk.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Natalia Valadares de Moraes (Other)
Collaborators: Hospital das Clínicas de Ribeirão Preto (Other)
Responsible Party: Sponsor-Investigator, Natalia Valadares de Moraes, Professor of Toxicology, Universidade Estadual Paulista Júlio de Mesquita Filho
Organization: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIFEDABCG2BCRP
Record Dates: First submitted 2018-07-17; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Drug Transporter
MeSH Terms: interventions — Blood Specimen Collection; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Wild homozygous for ABCG2 c.421C>A (Active Comparator): Chronic hypertensive breastfeeding women (18-45 years old) genotyped as wild homozygous for ABCG2 c.421C>A.
  Interventions: Procedure: Blood and breast milk sampling; Drug: Nifedipine
- Variant genotypes for ABCG2 c.421C>A (Experimental): Chronic hypertensive breastfeeding women (18-45 years old) genotyped as heterozygous or mutant homozygous for ABCG2 c.421C>A.
  Interventions: Procedure: Blood and breast milk sampling; Drug: Nifedipine

INTERVENTIONS:
Procedure: Blood and breast milk sampling — At least 15 days after starting treatment with 20 mg slow-release nifedipine every 12 hours. Blood and breast milk will be sampled before first dosing in the morning.
  Other Names: Biological samples for nifedipine analysis
Drug: Nifedipine — Chronic hypertensive breastfeeding women will be treated with slow-release 20 mg nifedipine, twice a day.
  Other Names: 20 mg nifedipine (slow-release)

SUMMARY:
This study aims to investigate the influence of the c.421C>A genetic polymorphism of the ABCG2 / BCRP transporter in the concentration ratio of nifedipine in maternal milk:plasma in hypertensive breastfeeding women attended at the Gynecology and Obstetrics Service of the Medical School of Ribeirão Preto, of the University of São Paulo. Thus, plasma and breast milk samples are being collected from patients in chronic use of the drug (n=30) within 15 to 30 days postnatal.

DETAILED DESCRIPTION:
The breast cancer resistance protein (ABCG2/BCRP) human transporter, encoded by the ABCG2 gene, is highly expressed on the human lactating breast. Nifedipine, a known substrate of ABCG2, is used for the treatment of hypertension in pregnancy and during breastfeeding. ABCG2 plays an important role on secreting drugs and xenobiotics into milk. The aim of the present study was to evaluate the effect of ABCG2 c.421C>A on nifedipine breast milk/plasma concentration ratio in hypertensive breastfeeding women. Nineteen hypertensive breastfeeding women treated with 20 mg slow-release nifedipine every 12 hours were investigated. Blood and breast milk samples were collected simultaneously 15-30 days after delivery and at least 15 days after drug treatment, in order to reach drug steady state. All patients were genotyped for ABCG2 c.421C>A using real time-PCR. Nifedipine concentration was determined in plasma and breast milk by high-performance liquid chromatography using UV detection. The comprehension of the variability in the transport of nifedipine to breast milk in hypertensive breastfeeding women will contribute to the evaluation of drug exposure in breast-fed infants to nifedipine and other ABCG2 substrates.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hypertensive breastfeeding women
* Patients being treated with 20 mg slow-release nifedipine every 12 hours for at least 15 days

Exclusion Criteria:

* Patients in use of ABCG2 inhibitors (omeprazole, pantoprazole, ritonavir, saquinavir, imatinib, efavirenz, nicardipine, abacavir, tacrolimus, ciclosporin A, cannabidiol);
* Patients who presented nifedipine adverse drug reactions
* Patients whose blood pressure normalized after delivery
* Patients who interrupted breastfeeding during the study
* Patients who did not return to the hospital for the clinical protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 19 (Estimated)
Dates: Start 2015-12-14 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Nifedipine concentration in plasma/milk ratio | After reaching steady state (at least 15 days of treatment), samples will be collected before first nifedipine dosing in the morning.
  The concentration ratio will be determined as (nifedipine concentration in plasma)/(nifedipine concentration in breast milk).

SECONDARY OUTCOMES:
Nifedipine concentration in plasma | After reaching steady state (at least 15 days of treatment), samples will be collected before first nifedipine dosing in the morning.
  The concentration of nifedipine in plasma determined by HPLC.
Nifedipine concentration in milk | After reaching steady state (at least 15 days of treatment), samples will be collected before first nifedipine dosing in the morning.
  The concentration of nifedipine in breast milk determined by HPLC.

IPD SHARING:
Plan to Share IPD: No